CLINICAL TRIAL: NCT00276484
Title: A Multicenter, Rand., Double-Blind, Titration Study to Evaluate & Compare the Efficacy & Safety of Ezetimibe Plus Atorvastatin Vs Atorvastatin in Hypercholesterolemic Pts. at High Risk for CHD Not Adequately Controlled on Atorvastatin 40 Mg
Brief Title: To Evaluate Ezetimibe Plus Atorvastatin Versus Atorvastatin in Patients With High Cholesterol Not Controlled on Atorvastatin 40 mg (0653-090)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0653-090; 2005_105
Record Dates: First submitted 2006-01-11; First posted 2006-01-13 (Estimated); Results first posted 2009-04-13 (Estimated); Last update posted 2024-05-14 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Atorvastatin; Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Active Comparator): Atorvastatin 80 mg
  Interventions: Drug: atorvastatin
- 2 (Experimental): Atorvastatin 40 mg + ezetimibe 10 mg
  Interventions: Drug: atorvastatin; Drug: ezetimibe

INTERVENTIONS:
Drug: atorvastatin — Atorvastatin 80 mg tablet by mouth, once a day for 6 weeks
  Arms: 1
Drug: atorvastatin — Atorvastatin 40 mg by mouth, once a day for 6 weeks
  Arms: 2
Drug: ezetimibe — Ezetimibe 10 mg tablets by mouth, once a day for 6 weeks.
  Arms: 2

SUMMARY:
To Evaluate and Compare the Efficacy and Safety of Ezetimibe Plus Atorvastatin Versus Atorvastatin in Hypercholesterolemic Patients at High Risk for Coronary Heart Disease Not Adequately Controlled on Atorvastatin 40 mg.

ELIGIBILITY:
Inclusion Criteria:

* Patient with LDL-C >70 mg/dL & on a stable dose of atorvastatin 40 mg

Exclusion Criteria:

* Pregnant or lactating women or intending to become pregnant
* Patient with sensitivity or intolerance to ezetimibe or atorvastatin

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 579 (Actual)
Dates: Start 2006-02; Primary Completion 2008-02 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leiter LA, Bays H, Conard S, Bird S, Rubino J, Hanson ME, Tomassini JE, Tershakovec AM. Efficacy and safety of ezetimibe added on to atorvastatin (40 mg) compared with uptitration of atorvastatin (to 80 mg) in hypercholesterolemic patients at high risk of coronary heart disease. Am J Cardiol. 2008 Dec 1;102(11):1495-501. doi: 10.1016/j.amjcard.2008.09.076. Epub 2008 Oct 23. PMID 19026303
- [Derived] Bays H, Conard S, Leiter LA, Bird S, Jensen E, Hanson ME, Shah A, Tershakovec AM. Are post-treatment low-density lipoprotein subclass pattern analyses potentially misleading? Lipids Health Dis. 2010 Nov 30;9:136. doi: 10.1186/1476-511X-9-136. PMID 21118495
- [Derived] Conard S, Bays H, Leiter LA, Bird S, Lin J, Hanson ME, Shah A, Tershakovec AM. Ezetimibe added to atorvastatin compared with doubling the atorvastatin dose in patients at high risk for coronary heart disease with diabetes mellitus, metabolic syndrome or neither. Diabetes Obes Metab. 2010 Mar;12(3):210-8. doi: 10.1111/j.1463-1326.2009.01152.x. PMID 20151997

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase III
  First Patient In: 4/6/2006; Last Patient Last Visit 2/26/2008
  96 centers worldwide (US, Canada)
  Eligible patients include those on a stable dose of atorvastatin 40 mg; or patients with adjusted LDLC
  pre-screen ranges who were treated with other lipid modifying therapy, or were statin and/or ezetimibe naïve.
Pre-assignment Details: Patients received and were blinded to atorvastatin 40 mg for a 4/5- week run-in period.
  Patients needed an LDL-C ≥ 70 mg/dL and ≤ 160 mg/dL at Visit 2 (week -1). Eligible patients were randomized at Visit 3 (Week 0) to either atorvastatin 80 mg or addition of ezetimibe 10 mg to their 40 mg dose of atorvastatin for a 6-week treatment period.
Groups:
- Atorvastatin + Ezetemibe: Atorvastatin 40 mg + Ezetemibe 10 mg every day for 6 weeks
- Atorvastatin: Atorvastatin 80 mg every day for 6 weeks
Period: Overall Study
Arm/Group | Atorvastatin + Ezetemibe | Atorvastatin
Started | 288 | 291
Completed | 279 | 278
Not Completed | 9 | 13
Not completed — Adverse Event | 4 | 7
Not completed — Lost to Follow-up | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Could not take time off work | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atorvastatin + Ezetemibe | Atorvastatin | Total
Number analyzed (Participants) | 288 | 291 | 579
Age, Continuous [Mean (Full Range); unit: years] | 60.6 [31 to 80] | 62 [34 to 79] | 61.3 [31 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 113 | 228
  Male | 173 | 178 | 351
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 237 | 232 | 469
  Asian | 4 | 8 | 12
  Black | 32 | 29 | 61
  Multi-Racial | 15 | 22 | 37
Apolipoprotein A-I [Mean (Standard Deviation); unit: mg/dL] | 154.0 (25.5) | 154.6 (25.0) | 154.3 (25.3)
Apolipoprotein B [Mean (Standard Deviation); unit: mg/dL] | 101.3 (19.0) | 102.0 (18.8) | 101.7 (18.9)
Apolipoprotein B:Apolipoprotein A-I ratio [Mean (Standard Deviation); unit: Ratio] | 0.7 (0.2) | 0.7 (0.2) | 0.7 (0.2)
C Reactive Protein [Mean (Standard Deviation); unit: mg/dL] | 1.8 (2.7) | 1.5 (3.0) | 1.6 (2.8)
High-Density Lipoprotein [Mean (Standard Deviation); unit: mg/dL] | 47.4 (10.5) | 47.2 (10.6) | 47.3 (10.5)
Low-Density Lipoprotein [Mean (Standard Deviation); unit: mg/dL] | 88.8 (16.2) | 89.8 (16.2) | 89.4 (16.2)
Low-Density Lipoprotein-C:High-Density Lipoprotein-C ratio [Mean (Standard Deviation); unit: Ratio] | 2.0 (0.6) | 2.0 (0.6) | 2.0 (0.6)
Non-High-Density Lipoprotein Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 117.7 (20.8) | 118.1 (21.9) | 117.9 (21.4)
Non-High-Density Lipoprotein-C:High-Density Lipoprotein-C ratio [Mean (Standard Deviation); unit: Ratio] | 2.6 (0.8) | 2.6 (0.8) | 2.6 (0.8)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 165.2 (21.4) | 165.3 (22.8) | 165.2 (22.1)
Total cholesterol:High-Density Lipoprotein-C ratio [Mean (Standard Deviation); unit: Ratio] | 3.6 (0.8) | 3.6 (0.8) | 3.6 (0.8)
Triglycerides [Median (Standard Deviation); unit: mg/dL] | 132.5 (72.1) | 134.0 (72.1) | 133.5 (72.1)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Week 6 in Low-Density Lipoprotein (LDL)-C
Description: Percent Change in LDL-C = [(week 6 value - baseline value)/baseline value]*100%
Time Frame: Baseline and 6 weeks
Population: Full Analysis Set (FAS): The FAS population includes all randomized patients who took at least 1 dose of study medication and had a baseline (BL) value and at least one post BL value. Post BL measurements up to 3 days following the last dose of double-blind study medication were included in the analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorvastatin + Ezetemibe | Atorvastatin
Number analyzed (Participants) | 277 | 279
Percent Change | -27.4 [-29.6 to -25.1] | -11.0 [-13.2 to -8.8]
Statistical Analysis 1: Comparison: Atorvastatin + Ezetemibe vs Atorvastatin; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment and baseline LDL-C value; Mean Difference (Final Values) = -16.3, 95% CI [-19.4 to -13.2], Standard Error of Mean 1.6

2. Secondary Outcome: Percent Change From Baseline to Week 6 in High-Density Lipoprotein Cholesterol (HDL-C)
Description: Percent Change in HDL-C = [(week 6 value - baseline value)/baseline value]*100%
Time Frame: Baseline and 6 weeks
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorvastatin + Ezetemibe | Atorvastatin
Number analyzed (Participants) | 277 | 279
Percent Change | -0.5 [-1.6 to 0.7] | -1.0 [-2.1 to 0.2]
Statistical Analysis 1: Comparison: Atorvastatin + Ezetemibe vs Atorvastatin; Test type: Superiority or Other; p = 0.551, ANCOVA; Model terms: treatment and baseline HDL-C value; Mean Difference (Final Values) = 0.5, 95% CI [-1.1 to 2.1], Standard Error of Mean 0.8

3. Secondary Outcome: Percent Change From Baseline to Week 6 in Non-High-Density Lipoprotein Cholesterol (Non-HDL-C)
Description: Percent Change in Non-HDL-C = [(week 6 value - baseline value)/baseline value]*100%
Time Frame: Baseline and 6 Weeks
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorvastatin + Ezetemibe | Atorvastatin
Number analyzed (Participants) | 277 | 279
Percent Change | -23.3 [-25.3 to -21.4] | -9.0 [-11.0 to -7.1]
Statistical Analysis 1: Comparison: Atorvastatin + Ezetemibe vs Atorvastatin; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment and baseline non-HDL-C value; Mean Difference (Final Values) = -14.3, 95% CI [-17.1 to -11.6], Standard Error of Mean 1.4

4. Secondary Outcome: Percent Change From Baseline to Week 6 in Total-Cholesterol
Description: Percent Change in Total-C = [(week 6 value - baseline value)/baseline value]*100%
Time Frame: Baseline and 6 Weeks
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorvastatin + Ezetemibe | Atorvastatin
Number analyzed (Participants) | 277 | 279
Percent Change | -16.9 [-18.3 to -15.4] | -6.9 [-8.4 to -5.5]
Statistical Analysis 1: Comparison: Atorvastatin + Ezetemibe vs Atorvastatin; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment and baseline Total-C value; Mean Difference (Final Values) = -10.0, 95% CI [-12.0 to -7.9], Standard Error of Mean 1.0

5. Secondary Outcome: Percent Change From Baseline to Week 6 in Triglycerides (TG)
Description: Percent Change in TG = [(week 6 value - baseline value)/baseline value]*100%
Time Frame: Baseline and 6 Weeks
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorvastatin + Ezetemibe | Atorvastatin
Number analyzed (Participants) | 277 | 279
Percent Change | -12.3 [-16.3 to -8.2] | -5.9 [-10.2 to -0.7]
Statistical Analysis 1: Comparison: Atorvastatin + Ezetemibe vs Atorvastatin; Test type: Superiority or Other; p < 0.001, Nonparametric ANCOVA; ANCOVA using ranks based on normal scores (Tukey method) with model terms for treatment and baseline triglycerides value; Median Difference (Final Values) = -7.3, 95% CI [-11.5 to -3.1] — The median difference is based on the Hodges-Lehmann estimates of shift; The distribution-free 95% CI is based on Wilcoxon's rank sum test statistic

6. Secondary Outcome: Percent Change From Baseline to Week 6 in Apolipoprotein B (Apo B)
Description: Percent Change in Apo B = [(week 6 value - baseline value)/baseline value]*100%
Time Frame: Baseline and 6 Weeks
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorvastatin + Ezetemibe | Atorvastatin
Number analyzed (Participants) | 275 | 276
Percent Change | -17.8 [-19.6 to -16.0] | -7.7 [-9.5 to -5.8]
Statistical Analysis 1: Comparison: Atorvastatin + Ezetemibe vs Atorvastatin; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment and baseline Apo B value; Mean Difference (Final Values) = -10.1, 95% CI [-12.7 to -7.6], Standard Error of Mean 1.3

7. Secondary Outcome: Percent Change From Baseline to Week 6 in Apolipoprotein A-I (Apo A-I)
Description: Percent Change in Apo A-I = [(week 6 value - baseline value)/baseline value]*100%
Time Frame: Baseline and 6 Weeks
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorvastatin + Ezetemibe | Atorvastatin
Number analyzed (Participants) | 275 | 276
Percent Change | -0.3 [-1.5 to 0.9] | -1.2 [-2.3 to -0.0]
Statistical Analysis 1: Comparison: Atorvastatin + Ezetemibe vs Atorvastatin; Test type: Superiority or Other; p = 0.313, ANCOVA; Model terms: treatment and baseline Apo A-I value; Mean Difference (Final Values) = 0.9, 95% CI [-0.8 to 2.5], Standard Error of Mean 0.8

8. Secondary Outcome: Percent Change From Baseline to Week 6 in Total-Cholesterol (TC):High-Density Lipoprotein Cholesterol (HDL-C) Ratio
Description: Percent Change in TC:HDL-C Ratio = [(week 6 ratio - baseline ratio)/baseline ratio]*100%
Time Frame: Baseline and 6 Weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorvastatin + Ezetemibe | Atorvastatin
Number analyzed (Participants) | 277 | 279
Percent Change | -16.0 [-176.6 to -14.4] | -5.6 [-7.2 to -4.1]
Statistical Analysis 1: Comparison: Atorvastatin + Ezetemibe vs Atorvastatin; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment and baseline Total-C:HDL-C value; Mean Difference (Final Values) = -10.4, 95% CI [-12.6 to -8.2], Standard Error of Mean 1.1

9. Secondary Outcome: Percent Change From Baseline to Week 6 in Low-Density Lipoprotein-Cholesterol:High-Density Lipoprotein-Cholesterol (LDL-C:HDL-C) Ratio
Description: Percent Change in LDL-C:HDL-C Ratio = [(week 6 ratio - baseline ratio)/baseline ratio]*100%
Time Frame: Baseline and 6 Weeks
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Atorvastatin + Ezetemibe | Atorvastatin
Number analyzed (Participants) | 277 | 279
Percent change | -26.4 [-28.8 to -24.0] | -9.9 [-12.3 to -7.5]
Statistical Analysis 1: Comparison: Atorvastatin + Ezetemibe vs Atorvastatin; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment and baseline LDL-C:HDL-C value; Mean Difference (Final Values) = -16.5, 95% CI [-19.9 to -13.1], Standard Error of Mean 1.7

10. Secondary Outcome: Percent Change From Baseline to Week 6 in Apolipoprotein B:Apolipoprotein A-I (Apo B:Apo A-I) Ratio
Description: Percent Change in Apo B:Apo A-I Ratio = [(week 6 ratio - baseline ratio)/baseline ratio]*100%
Time Frame: Baseline and 6 Weeks
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorvastatin + Ezetemibe | Atorvastatin
Number analyzed (Participants) | 275 | 276
Percent Change | -16.9 [-18.9 to -14.9] | -5.9 [-7.9 to -3.9]
Statistical Analysis 1: Comparison: Atorvastatin + Ezetemibe vs Atorvastatin; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment and baseline Apo B:Apo A-I value; Mean Difference (Final Values) = -11.0, 95% CI [-13.8 to -8.2], Standard Error of Mean 1.4

11. Secondary Outcome: Percent Change From Baseline to Week 6 in Non-High-Density Lipoprotein-Cholesterol:High-Density Lipoprotein-Cholesterol (Non-HDL-C:HDL-C) Ratio
Description: Percent Change in non-HDL-C:HDL-C Ratio = [(week 6 ratio - baseline ratio)/baseline ratio]*100%
Time Frame: Baseline and 6 Weeks
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorvastatin + Ezetemibe | Atorvastatin
Number analyzed (Participants) | 277 | 279
Percent Change | -22.2 [-24.5 to -19.9] | -7.6 [-9.9 to -5.4]
Statistical Analysis 1: Comparison: Atorvastatin + Ezetemibe vs Atorvastatin; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment and baseline non-HDL-C:HDL-C value; Mean Difference (Final Values) = -14.5, 95% CI [-17.7 to -11.3], Standard Error of Mean -1.6

12. Secondary Outcome: Percent Change From Baseline to Week 6 in C Reactive Protein (CRP)
Description: Percent Change in CRP = [(week 6 value - baseline value)/baseline value]*100%
Time Frame: Baseline and 6 Weeks
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Atorvastatin + Ezetemibe | Atorvastatin
Number analyzed (Participants) | 277 | 276
Percent Change | -18.3 [-25.0 to -11.1] | -11.5 [-18.7 to -3.6]
Statistical Analysis 1: Comparison: Atorvastatin + Ezetemibe vs Atorvastatin; Test type: Superiority or Other; p = 0.174, Longitudinal Data Analysis (LDA); LDA method of Liang and Zeger with model terms: treatment, time, and the interaction of time by treatment; Mean Difference (Final Values) = -6.8, 95% CI [-17.1 to 3.4] — Data for analysis was transformed by the natural log and the difference in geometric mean % change from BL calculated based on the difference in the back-transformed least squares means

13. Secondary Outcome: Number of Patients Who Attained Target Low-Density Lipoprotein Cholesterol (LDL-C) <70 mg/dL at Week 6
Time Frame: 6 Weeks
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Atorvastatin + Ezetemibe | Atorvastatin
Number analyzed (Participants) | 277 | 279
Participants
  <70 mg/dL | 204 | 88
  >=70 mg/dL | 73 | 191
Statistical Analysis 1: Comparison: Atorvastatin + Ezetemibe vs Atorvastatin; Test type: Superiority or Other; p < 0.001, Regression, Logistic; Model terms: treatment and baseline LDL-C value; Odds Ratio (OR) = 8.37, 95% CI [5.45 to 12.84]

ADVERSE EVENTS:
Arm/Group | Atorvastatin + Ezetemibe | Atorvastatin
Serious Adverse Events (participants affected / at risk) | 9 | 5
Other Adverse Events (participants affected / at risk) | 63 | 61
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Atorvastatin + Ezetemibe | Atorvastatin
Anaemia (Blood and lymphatic system disorders) | 0/286 | 1/289
Cardiac failure congestive (Cardiac disorders) | 1/286 | 0/289
Coronary artery disease (Cardiac disorders) | 0/286 | 1/289
Myocardial infarction (Cardiac disorders) | 3/286 | 1/289
Gastritis (Gastrointestinal disorders) | 0/286 | 1/289
Chest pain (General disorders) | 1/286 | 0/289
Hernia obstructive (General disorders) | 0/286 | 1/289
Non-cardiac chest pain (General disorders) | 1/286 | 0/289
Pneumonia (Infections and infestations) | 1/286 | 0/289
Overdose (Injury, poisoning and procedural complications) | 0/286 | 1/289
Presyncope (Nervous system disorders) | 1/286 | 0/289
Mental status (Psychiatric disorders) | 0/286 | 1/289
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1/286 | 0/289
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1/286 | 0/289
Hypertensive crisis (Vascular disorders) | 1/286 | 0/289
Labile hypertension (Vascular disorders) | 1/286 | 0/289
Peripheral vascular disorder (Vascular disorders) | 0/286 | 1/289
OTHER ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Atorvastatin + Ezetemibe | Atorvastatin
Anaemia (Blood and lymphatic system disorders) | 1/286 | 1/289
Cardiac failure congestive (Cardiac disorders) | 1/286 | 0/289
Coronary artery disease (Cardiac disorders) | 0/286 | 1/289
Myocardial infarction (Cardiac disorders) | 3/286 | 1/289
Vertigo (Ear and labyrinth disorders) | 1/286 | 0/289
Retinal detachment (Eye disorders) | 1/286 | 0/289
Vision blurred (Eye disorders) | 2/286 | 1/289
Visual disturbance (Eye disorders) | 0/286 | 1/289
Abdominal discomfort (Gastrointestinal disorders) | 0/286 | 1/289
Abdominal distension (Gastrointestinal disorders) | 0/286 | 1/289
Abdominal pain (Gastrointestinal disorders) | 2/286 | 2/289
Abdominal pain upper (Gastrointestinal disorders) | 0/286 | 1/289
Constipation (Gastrointestinal disorders) | 1/286 | 2/289
Dental caries (Gastrointestinal disorders) | 1/286 | 0/289
Diarrhoea (Gastrointestinal disorders) | 0/286 | 6/289
Diverticulum (Gastrointestinal disorders) | 1/286 | 0/289
Dyspepsia (Gastrointestinal disorders) | 0/286 | 2/289
Dysphagia (Gastrointestinal disorders) | 1/286 | 0/289
Flatulence (Gastrointestinal disorders) | 1/286 | 0/289
Gastritis (Gastrointestinal disorders) | 0/286 | 1/289
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1/286 | 0/289
Gingivitis (Gastrointestinal disorders) | 1/286 | 0/289
Nausea (Gastrointestinal disorders) | 2/286 | 2/289
Stomach discomfort (Gastrointestinal disorders) | 1/286 | 1/289
Vomiting (Gastrointestinal disorders) | 1/286 | 1/289
Chest pain (General disorders) | 3/286 | 2/289
Fatigue (General disorders) | 0/286 | 4/289
Hernia obstructive (General disorders) | 0/286 | 1/289
Non-cardiac chest pain (General disorders) | 1/286 | 0/289
Oedema peripheral (General disorders) | 2/286 | 1/289
Pyrexia (General disorders) | 0/286 | 1/289
Cholelithiasis (Hepatobiliary disorders) | 1/286 | 0/289
Seasonal allergy (Immune system disorders) | 1/286 | 1/289
Bronchitis (Infections and infestations) | 4/286 | 1/289
Chronic sinusitis (Infections and infestations) | 1/286 | 0/289
Conjunctivitis infective (Infections and infestations) | 0/286 | 1/289
Gastroenteritis viral (Infections and infestations) | 0/286 | 1/289
Nasopharyngitis (Infections and infestations) | 4/286 | 1/289
Pharyngitis (Infections and infestations) | 0/286 | 1/289
Pharyngitis streptococcal (Infections and infestations) | 0/286 | 1/289
Pneumonia (Infections and infestations) | 1/286 | 0/289
Sinusitis (Infections and infestations) | 2/286 | 1/289
Upper respiratory tract infection (Infections and infestations) | 1/286 | 7/289
Urinary tract infection (Infections and infestations) | 0/286 | 1/289
Back injury (Injury, poisoning and procedural complications) | 1/286 | 0/289
Burns second degree (Injury, poisoning and procedural complications) | 1/286 | 0/289
Contusion (Injury, poisoning and procedural complications) | 2/286 | 0/289
Joint sprain (Injury, poisoning and procedural complications) | 0/286 | 1/289
Overdose (Injury, poisoning and procedural complications) | 0/286 | 1/289
Scratch (Injury, poisoning and procedural complications) | 0/286 | 1/289
Thermal burn (Injury, poisoning and procedural complications) | 1/286 | 0/289
Tooth fracture (Injury, poisoning and procedural complications) | 1/286 | 0/289
Alanine aminotransferase (General disorders) | 2/286 | 2/289
Aspartate aminotransferase (General disorders) | 2/286 | 2/289
Blood bilirubin increased (General disorders) | 0/286 | 1/289
Blood creatine phosphokinase increased (General disorders) | 2/286 | 0/289
Blood potassium increased (General disorders) | 2/286 | 0/289
Blood uric acid increased (General disorders) | 1/286 | 0/289
Carotid pulse decreased (General disorders) | 1/286 | 0/289
Gamma-glutamyltransferase increased (General disorders) | 2/286 | 1/289
Arthralgia (Musculoskeletal and connective tissue disorders) | 0/286 | 4/289
Back pain (Musculoskeletal and connective tissue disorders) | 0/286 | 3/289
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1/286 | 0/289
Joint effusion (Musculoskeletal and connective tissue disorders) | 1/286 | 0/289
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0/286 | 2/289
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1/286 | 0/289
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0/286 | 1/289
Myalgia (Musculoskeletal and connective tissue disorders) | 1/286 | 5/289
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4/286 | 3/289
Carotid artery stenosis (Nervous system disorders) | 0/286 | 1/289
Cerebellar ataxia (Nervous system disorders) | 1/286 | 0/289
Dizziness (Nervous system disorders) | 3/286 | 2/289
Headache (Nervous system disorders) | 4/286 | 2/289
Migraine (Nervous system disorders) | 1/286 | 0/289
Paraesthesia (Nervous system disorders) | 1/286 | 0/289
Presyncope (Nervous system disorders) | 1/286 | 0/289
Sciatica (Nervous system disorders) | 0/286 | 1/289
Syncope (Nervous system disorders) | 1/286 | 0/289
Anxiety (Psychiatric disorders) | 1/286 | 1/289
Confusional state (Psychiatric disorders) | 1/286 | 0/289
Insomnia (Psychiatric disorders) | 0/286 | 1/289
Mental status changes (Psychiatric disorders) | 0/286 | 1/289
Calculus bladder (Renal and urinary disorders) | 0/286 | 1/289
Nephrolithiasis (Renal and urinary disorders) | 1/286 | 0/289
Renal cyst (Renal and urinary disorders) | 1/286 | 0/289
Renal failure (Renal and urinary disorders) | 1/286 | 0/289
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1/286 | 1/289
Erectile dysfunction (Reproductive system and breast disorders) | 0/286 | 1/289
Asthma (Respiratory, thoracic and mediastinal disorders) | 0/286 | 1/289
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1/286 | 0/289
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1/286 | 1/289
Cough (Respiratory, thoracic and mediastinal disorders) | 0/286 | 1/289
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3/286 | 1/289
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0/286 | 1/289
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1/286 | 0/289
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1/286 | 0/289
Pruritus (Skin and subcutaneous tissue disorders) | 1/286 | 1/289
Rash erythematous (Skin and subcutaneous tissue disorders) | 0/286 | 1/289
Cataract operation (General disorders) | 0/286 | 1/289
Inguinal hernia repair (General disorders) | 1/286 | 0/289
Haematoma (Vascular disorders) | 0/286 | 1/289
Hypertension (Vascular disorders) | 1/286 | 0/289
Hypertensive crisis (Vascular disorders) | 1/286 | 0/289
Hypotension (Vascular disorders) | 1/286 | 0/289
Labile hypertension (Vascular disorders) | 1/286 | 0/289
Peripheral vascular disorder (Vascular disorders) | 0/286 | 1/289

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.